CLINICAL TRIAL: NCT01968525
Title: The Effect of Chronic Anemia on Safety Period of Tracheal Intubation in Gynecology Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Geng guiqi, PhD, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 199987
Record Dates: First submitted 2013-10-12; First posted 2013-10-24 (Estimated); Last update posted 2013-10-24 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Anemia
Keywords: anemia; non-hypoxic apnoea; tracheal intubation; anesthesia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group A (Experimental): the hemoglobin is >12g/L in patients from group A.
  Interventions: Biological: pre-oxygen
- Group B (Experimental): Hb 9-12g/L
  Interventions: Biological: pre-oxygen
- Group C (Experimental): Hb<9g/L
  Interventions: Biological: pre-oxygen

INTERVENTIONS:
Biological: pre-oxygen — 3 min of preoxygenation before anesthesia induction.

SUMMARY:
1. Every individual receiving a general anesthetic is at potential risk for developing a ''cannot intubate-cannot ventilate'' situation following anesthetic induction.
2. Building up of oxygen reserves assumes great significance as this provides a longer duration of non-hypoxic apnea should one be faced with an unanticipated difficult airway.
3. The main physiological functions of red blood cell hemoglobin are to deliver oxygen to the peripheral tissues.
4. During anemia, a reduction in blood oxygen content occurs as a result of reduced Hb while arterial oxygenation and oxyhemoglobin saturation remain high.
5. Previous studies about the duration of non-hypoxic apnoea focus on methods to improve the safety period of tracheal intubation.
6. To our knowledge, there is no literature about the duration of non-hypoxic apnoea of anemia patients.
7. The aim of this study was to assess the effect of chronic anemia on the duration of non-hypoxic apnoea during induction of anaesthesia.

DETAILED DESCRIPTION:
After breathing for 3 minutes, anesthesia induction was conducted. The endotracheal tube position was confirmed after anesthesia induction. Patients were left apneic with the endotracheal tube open to room air. The non-hypoxic apneic period was recorded as the time (in seconds) taken for the drop in pulse saturation to 90% or an apneic period of 10 min elapsed, whichever was earlier.

ELIGIBILITY:
Inclusion Criteria:

1. patients scheduled to undergo general anesthesia
2. American Society of Anesthesiologists Performance Status 1-2
3. adults

Exclusion Criteria:

1. Individuals with significant cardiorespiratory or cerebrovascular disease,
2. difficult intubation
3. history of epilepsy
4. body mass index >25 kg/m2,
5. and those who had smoking history in past 6 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2013-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
duration of non-hypoxic apnoea | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Guiqi Geng, PhD, Study Director — Department of anesthesiology, obstetrics and genecology hospital, FuDan university
Locations (1):
- Fudan university, Shanghai, Shanghai Municipality, China